CLINICAL TRIAL: NCT00982891
Title: Palliation of Dyspnea in Advanced Chronic Obstructive Pulmonary Disease: Understanding Patients' and Caregivers' Experiences of Opioid Therapy
Brief Title: Palliation of Dyspnea in Advanced Chronic Obstructive Pulmonary Disease (COPD)
Acronym: ROS-003
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Nova Scotia Health Research Foundation (Other Government); Atlantic Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Graeme Rocker, Professor of Medicine, Nova Scotia Health Authority
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ROS-003; CIHR IHP 94532
Record Dates: First submitted 2009-09-21; First posted 2009-09-23 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: chronic obstructive pulmonary disease; palliation; opioids
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Analgesics, Opioid; Morphine; Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Morphine, low dose, in addition to conventional treatment (Experimental): Morphine dose titration
  Interventions: Drug: Opioid (morphine sulphate) in low dose

INTERVENTIONS:
Drug: Opioid (morphine sulphate) in low dose — individualized titration
  Other Names: M-ESLON (DIN 02019930); morphine sulphate (SR); Doloral 1 (DIN 00614491); morphine hydrochloride; Doloral 5 (DIN 00614505); pms-Hydromorphone (DIN 01916386); hydromorphone hydrochloride; Hydromorph Contin (DIN 02125323) - hydromorphone hydrochloride (SR)

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) affects at least 750,000 Canadians and is currently the 4th leading cause of death in Canada. Almost everyone with COPD suffers from shortness of breath (dyspnea) that worsens over time despite standard treatment (inhalers, exercise programs and oxygen). Patients and families have identified relief from dyspnea as a top priority for improved care. New approaches are needed for treating advanced COPD to lessen the burden that it places on the lives of patients and families alike. Opioid drugs, such as morphine, can help in COPD in many ways, including reducing dyspnea, fear and anxiety. Opioids are used widely in cancer for similar symptoms. However, there are historical biases against their use in advanced COPD (mostly due to fear of side effects when much higher doses than the investigators intend have been used in the past). No studies have assessed the value to patients of using low dose opioids in advanced COPD in addition to conventional treatment. The investigators are planning a study that involves recording interviews with about 30 patients and their partner or key family member before and after starting treatment with low dose morphine, to understand their experiences with using morphine. The investigators will also ask them to complete questionnaires about quality of life, dyspnea, anxiety, depression and fear. Descriptions of experiences of using morphine have the potential to inform patients, families, clinicians and professional societies about the benefits and harms of opioid use for dyspnea in the advanced stages of a common serious lung disease when traditional treatments often fail. The investigators will conduct the study in both urban (Halifax and Saskatoon) and in a rural setting (New Brunswick). The investigators' study of an inexpensive and widely available treatment has the potential to improve care and outcomes in advanced COPD for the many Canadians living and dying with this serious lung disease.

ELIGIBILITY:
Inclusion Criteria:

* We define advanced COPD as including those with severe COPD by CTS criteria (i.e., severe shortness of breath resulting in the patient being too breathless to leave the house, or breathlessness after dressing/undressing (i.e., Medical Research Council (MRC) score of 5), or the presence of chronic respiratory failure (PaCO2>45) or clinical signs of right heart failure).
* We will also include patients who are short of breath and stop walking after about 100 meters or a few minutes on the level (MRC score 4) with at least one the following:

  * BMI < 21;
  * post-bronchodilator FEV1 < 30% predicted;
  * one or more hospital admissions for acute exacerbation of COPD in the previous year.
* MRC 4 patients will be recruited only if their baseline Chronic Respiratory Questionnaire - dyspnea domain (CRQ-D) score is < 5, an entry criterion used in a Canadian RCT involving patients with advanced lung disease.

Exclusion Criteria:

* Patients and/or caregivers with cognitive or other difficulties that would preclude questionnaire completion.
* Inability to speak or understand English.
* Patients considered to be dying or with an expected survival of less than 2 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To understand the experiences of patients and informal caregivers living with severe COPD, following the addition of opioid therapy to conventional treatment. | 6 months

SECONDARY OUTCOMES:
To explore the effect of opioid therapy on dyspnea and on quality of life, anxiety, depression, caregiver experiences and to determine proportion of patients finding opioids helpful at 4-6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Graeme M Rocker, DM MHSc, Principal Investigator — Dalhousie University/QE II Health Sciences Centre, Halifax, NS
Locations (3):
- Canada (3):
  - Horizon Health Network, Saint John, New Brunswick
  - Capital District Health Authority, Halifax, Nova Scotia
  - Royal University Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Rocker GM, Simpson AC; Joanne Young BHSc; Horton R, Sinuff T, Demmons J; Margaret Donahue MDiv MAHSR; Hernandez P, Marciniuk D. Opioid therapy for refractory dyspnea in patients with advanced chronic obstructive pulmonary disease: patients' experiences and outcomes. CMAJ Open. 2013 Jan 24;1(1):E27-36. doi: 10.9778/cmajo.20120031. eCollection 2013 Jan. PMID 25077099